CLINICAL TRIAL: NCT05844345
Title: The Effect of Hydrocolloid Tape and Facial Massage on Nasal Injury, Comfort and Stress in Premature Infants During Noninvasive Mechanical Ventilation
Brief Title: The Effect of Hydrocolloid Tape and Facial Massage in Premature Infants During Noninvasive Mechanical Ventilation
Acronym: NIPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dilek Kucuk Alemdar, Associate professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KAEK39
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Nasal Injury
Keywords: nasal injury; hydrocolloid tape; non-invasive mechanical ventilation; premature; facial massage; stress; comfort
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental
Who Masked: Participant, Outcomes Assessor
Masking Description: After the preterm neonates abiding by the inclusion criteria in the research are randomly allocated to the study groups, parents will provide written consent with an informed volunteer consent form without giving parents information about which group their infant will be included in. The researcher will apply the hydrocolloid barrier and facial massage themselves, so the researcher will not be blinded. However, to prevent bias, research outcome measures will be recorded by two nurses who are employed in the NICU, are university graduates and who do not know which infant is in the experiment or control groups. With the aim of preventing bias during analysis of data, the database for the study groups will be coded A, B and C by someone other than the researcher, and analysis of data will be performed by an independent statistical expert. Blinding of outcome measures, statistical analysis and reporting will be performed with the aim of preventing statistical and reporting bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydrocolloid barrier group (Experimental): Premature infants will firstly be assessed by two nurses with undergraduate degrees working in the clinic in terms of neonatal skin condition score, nasal injury score, neonatal stress level and comfort score before beginning NIMV support. The colloid tape will be cut to a t-shape to cover across the bridge of the nose and the nasal septum and philtrum and placed on the infant's face.
  Interventions: Other: Hydrocolloid barrier group
- Facial Massage group (Experimental): Premature infants will firstly be assessed by two nurses with undergraduate degrees working in the clinic in terms of neonatal skin condition score, nasal injury score, neonatal stress level and comfort score before beginning NIMV support. After beginning NIMV support, the researcher will perform facial massage 2 times in each 12-hour shift.
  Interventions: Other: Facial Massage group
- Control group (No Intervention): Premature infants will firstly be assessed by two nurses with undergraduate degrees working in the clinic in terms of neonatal skin condition score, nasal injury score, neonatal stress level and comfort score before beginning NIMV support. After beginning NIMV support, no procedure apart from routine care will be performed. Routine care includes feeding every 3 hours, diaper care, position changes, changing the placement of probes and electrodes and confirming the position of the nasal cannula.

INTERVENTIONS:
Other: Hydrocolloid barrier group — In the hydrocolloid barrier group, Comfeel Plus brand hydrocolloid tape will be used. Hydrocolloid tape is a dressing cover made of soft, flexible and economic material in the form of a semi-permeable film or foam-supported gel. Air exchange continues due to the semipermeable film on the top, while entry of harmful microorganisms to the region is prevented, healing is accelerated by creating a humid environment for the wound and exudate from the wound is absorbed. These features reduce the risk of developing infection and ensure patient comfort. There is no specific change time, though generally the tape is changed every 3-5 days; however, it may remain in place for up to 7 days.
  Arms: Hydrocolloid barrier group
Other: Facial Massage group — Premature infants in the facial massage group will have facial massage applied by the researcher. For facial massage, physiological serum used for routine moisturizing in the clinic will be used. When performing facial massage, the fingers will be placed in the middle of the infant's forehead and massage will be performed towards the temples. The eyelids will be lightly rubbed toward the temples. Both thumbs will be placed in the center of the eyebrows and the ridge of the nose will be rubbed toward the lips. The sides of the nose will be rubbed with light pressure. The nasal septum will be rubbed toward the tip of the nose along the philtrum. The fingers will be placed on the philtrum region above the gums and the mouth will be rubbed toward the ears to make a smiling expression. The chin will be lightly massaged toward the back of the ears. The thumbs of both hands will rub from under the infant's chin toward the temples to give make a smiling face (smiling motion).
  Arms: Facial Massage group

SUMMARY:
The aim of this study is to assess the effect of nasal injury prevention interventions (NIPI) (hydrocolloid tape and facial massage) on nasal septum injury, stress and comfort of premature neonates (28-35 weeks gestation) receiving non-invasive mechanical ventilation (NIMV) support.

DETAILED DESCRIPTION:
The aim of this study is to assess the effect of nasal injury prevention interventions (NIPI) (hydrocolloid tape and facial massage) on nasal septum injury, stress and comfort of premature neonates receiving non-invasive mechanical ventilation (NIMV) support.

This study is a, prospective randomized controlled trial. The population for the research will comprise 108 premature neonates from 28-35 weeks gestation receiving NIMV support in the neonatal intensive care unit (NICU) from March 2023 to March 2024. Participants will be randomly assigned to one of three groups; the first group (n=40) will have hydrocolloid tape applied, the second group (n=40) will have facial massage and the third group (n=40 will be the control group. Research data will be collected with the Neonatal Descriptive Information Form, Nasal Injury Score Table (NIST), Neonate Skin Condition Scale (NSCS), Premature Infant Comfort Scale (COMFORT) and Neonatal Stress Scale (NSS).

Intervention Tools:

The NICU where the study will be performed uses SLEE 2000 and SLEE 5000 model mechanical ventilators. Both mechanical ventilators have no difference in implementation modes for invasive and non-invasive mechanical ventilation for term and premature infants. All premature infants included in the study will have NIMV support provided using SLEE 2000 and SLEE 5000 model mechanical ventilators. For NIMV of premature infants, NeoSmart brand (Mediplast Respiratory Products Sdn. Bhd, Malaysia) nasal cannulas will be used. The nasal cannula has soft binasal prongs and suitable structure for low- and high-flow oxygen use. A new sterile cannula will be used for each infant. There are 5 different sizes of x small, small, medium, large and x large. The sizes most frequently used for premature infants are small and medium.

In the hydrocolloid barrier group, Comfeel Plus brand hydrocolloid tape will be used. Hydrocolloid tape is a dressing cover made of soft, flexible and economic material in the form of a semi-permeable film or foam-supported gel (Başara, 2022; Ribeiro et al., 2020; Imbulana et al., 2018). Air exchange continues due to the semipermeable film on the top, while entry of harmful microorganisms to the region is prevented, healing is accelerated by creating a humid environment for the wound and exudate from the wound is absorbed. These features reduce the risk of developing infection and ensure patient comfort (Başara, 2022; Ribeiro et al., 2020; Imbulana et al., 2018; Fletcher et al. 2011; Xie, 2014). There is no specific change time, though generally the tape is changed every 3-5 days; however, it may remain in place for up to 7 days (Ribeiro et al., 2020; Fletcher et al. 2011).

Premature infants in the facial massage group will have facial massage applied by the researcher. The researcher has completed 120 hours of theoretical and practical training about infant massage and received the Infant Massage Certificate. For facial massage, physiological serum used for routine moisturizing in the clinic will be used. When performing facial massage, the fingers will be placed in the middle of the infant's forehead and massage will be performed towards the temples. The eyelids will be lightly rubbed toward the temples. Both thumbs will be placed in the center of the eyebrows and the ridge of the nose will be rubbed toward the lips. The sides of the nose will be rubbed with light pressure. The nasal septum will be rubbed toward the tip of the nose along the philtrum. The fingers will be placed on the philtrum region above the gums and the mouth will be rubbed toward the ears to make a smiling expression. The chin will be lightly massaged toward the back of the ears. The thumbs of both hands will rub from under the infant's chin toward the temples to give make a smiling face (smiling motion).

Hydrocolloid barrier group: Premature infants will firstly be assessed by two nurses with undergraduate degrees working in the clinic in terms of neonatal skin condition score, nasal injury score, neonatal stress level and comfort score before beginning NIMV support. The colloid tape will be cut to a t-shape to cover across the bridge of the nose and the nasal septum and philtrum and placed on the infant's face. For 3 days after beginning NIMV support, the same two nurses will assess the neonatal skin condition score, nasal injury score, neonatal stress level and comfort score at 24-hour intervals.

Facial Massage group: Premature infants will firstly be assessed by two nurses with undergraduate degrees working in the clinic in terms of neonatal skin condition score, nasal injury score, neonatal stress level and comfort score before beginning NIMV support. After beginning NIMV support, the researcher will perform facial massage 2 times in each 12-hour shift. For 3 days after beginning NIMV support, the same two nurses will assess the neonatal skin condition score, nasal injury score, neonatal stress level and comfort score at 24-hour intervals.

Control group: Premature infants will firstly be assessed by two nurses with undergraduate degrees working in the clinic in terms of neonatal skin condition score, nasal injury score, neonatal stress level and comfort score before beginning NIMV support. After beginning NIMV support, no procedure apart from routine care will be performed. Routine care includes feeding every 3 hours, diaper care, position changes, changing the placement of probes and electrodes and confirming the position of the nasal cannula. For 3 days after beginning NIMV support, the same two nurses will assess the neonatal skin condition score, nasal injury score, neonatal stress level and comfort score at 24-hour intervals. If nasal injury develops in the control group, antibacterial creams may be used in line with permission from the clinical doctor.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates between 28-34 weeks gestation,
* Preterm neonates beginning nasal NIMV due to respiratory distress within the first six hours after birth,
* Preterm neonates with nasal NIMV after invasive mechanical ventilation,
* Preterm neonates with parental consent to participate in the study.

Exclusion Criteria:

* Preterm neonates with congenital anomaly (choanal atresia, cleft palate-lip, esophagus atresia, tracheoesophageal fistula, etc.),
* Preterm neonates beginning NIMV support after more than 24 hours,
* Preterm neonates with skin diseases (ichthyosis, etc.),
* Preterm neonates with pulmonary hypertension.

Ages: 28 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Nasal Injury Score Table | 3 days
  The nasal injury score table was developed and was designed with the aim of assessing nasal injury in neonates receiving NIMV support. Pressure injury forming in 6 different anatomical regions of the nose is assessed from 0-4 points and the total points are obtained.
Neonatal Skin Condition Score | 3 days
  This is a 3-item scale developed to assess the dryness and presence and degree of erythema and disruption/peeling of the skin in preterm, term and post-term infants admitted to the NICU.

SECONDARY OUTCOMES:
Neonatal Stress Scale | every 12-hour shift over 3 days for assessment.
  With the aim of assessing stress in neonates, the validity and reliability for the scale was examined. The scale with 3-point Likert rating comprises a total of 24 items.
COMFORT scale | every 12-hour shift over 3 days for assessment.
  Premature infants with gestational age ≥28 and ≤37 weeks. The Turkish validity and reliability of the scale was examined.The scale with 5-point Likert rating assesses 7 parameters of consciousness, calmness/agitation, respiratory status or crying, physical movements, muscle tone, facial movements and mean heart rate. Each item is given points from bad to good of 1 to 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Dilek alemdar, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No